CLINICAL TRIAL: NCT07340866
Title: Physical Fatigue, Compassion Fatigue, and Quiet Quitting Tendency Among Physiotherapists in Türkiye: A Cross-Sectional Study
Brief Title: Physical Fatigue, Compassion Fatigue, and Quiet Quitting in Physiotherapists
Status: Not yet recruiting | Type: Observational
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, Mahmut Sürmeli, Assistant Professor, Tokat Gaziosmanpasa University
Other Study IDs: GOP-FTR-01-2025
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Quiet Quitting; Fatigue, Compassion; Work Engagement
Keywords: fatigue; compassion fatigue; work engagement; occupational health; quiet quitting
MeSH Terms: conditions — Compassion Fatigue; Fatigue | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Physiotherapists: Physiotherapists actively working in public or private healthcare institutions in Türkiye who voluntarily participate in the study.
  Interventions: Other: No Intervention (Observational Study)

INTERVENTIONS:
Other: No Intervention (Observational Study) — This is an observational study. No intervention is administered. Data are collected using self-report questionnaires.

SUMMARY:
Physiotherapists are exposed to both physical and emotional demands due to the nature of their profession. Repetitive physical workload, prolonged standing, patient handling, and continuous interaction with patients may contribute to physical fatigue and compassion fatigue. These factors may negatively affect work engagement and lead to a phenomenon known as quiet quitting, which refers to reduced psychological involvement in work without formally leaving the job.

The aim of this study is to examine levels of physical fatigue and compassion fatigue among physiotherapists working in Türkiye and to investigate their association with quiet quitting tendencies. This observational, cross-sectional study will include physiotherapists actively working in public or private healthcare settings. Data will be collected using validated self-report questionnaires administered online and face-to-face.

Understanding the relationship between occupational fatigue and quiet quitting may help inform strategies to improve well-being, job satisfaction, and sustainability in the physiotherapy workforce.

DETAILED DESCRIPTION:
Physiotherapists perform physically demanding tasks such as repetitive movements, patient transfers, and prolonged standing, while also managing emotional demands related to continuous patient care. These occupational stressors may lead to physical fatigue and compassion fatigue, which can negatively influence professional engagement and work sustainability. In recent years, the concept of quiet quitting has emerged to describe a reduction in psychological commitment to work while remaining formally employed. However, limited evidence exists regarding the relationship between occupational fatigue and quiet quitting among physiotherapists.

This study is designed as an observational, cross-sectional investigation aiming to evaluate physical fatigue, compassion fatigue, and quiet quitting tendencies among physiotherapists working in Türkiye. Eligible participants will be physiotherapists who have graduated from a Physiotherapy and Rehabilitation undergraduate program and are actively working in public or private healthcare institutions. Participation will be voluntary, and informed consent will be obtained electronically prior to data collection.

Data will be collected through face-to-face interviews and online platforms, including electronic survey tools and professional communication channels. Participants will complete a demographic and occupational information form followed by validated measurement instruments assessing compassion fatigue, physical fatigue, work-related musculoskeletal discomfort, and quiet quitting attitudes.

Statistical analyses will be conducted using appropriate descriptive and inferential methods. Relationships between variables will be examined using correlation analyses, and the predictive effects of physical fatigue and compassion fatigue on quiet quitting tendencies will be evaluated using multiple regression analysis. The findings of this study are expected to contribute to a better understanding of occupational well-being among physiotherapists and to provide evidence to support strategies aimed at improving working conditions and professional sustainability in rehabilitation services.

ELIGIBILITY:
Inclusion Criteria:

* Graduated from a Physiotherapy and Rehabilitation undergraduate program
* Actively working as a physiotherapist in Türkiye
* Voluntary participation and provision of informed consent

Exclusion Criteria:

* Refusal to participate in the study
* Working in a profession other than physiotherapy
* Incomplete or incorrectly completed questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of physiotherapists actively working in public or private healthcare institutions in Türkiye.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-22 (Estimated); Primary Completion 2026-04-23 (Estimated); Study Completion 2026-05-12 (Estimated)

PRIMARY OUTCOMES:
Quiet Quitting Tendency | At enrollment (single assessment)
  Quiet quitting tendency will be assessed using the Quiet Quitting Attitude Scale, a validated self-report questionnaire measuring reduced psychological engagement with work. Higher scores indicate a greater tendency toward quiet quitting.

SECONDARY OUTCOMES:
Physical Fatigue Level | At enrollment (single assessment)
  Physical fatigue will be assessed using the Fatigue Assessment Scale, a validated self-report measure evaluating physical and cognitive aspects of fatigue. Higher scores reflect greater fatigue severity.
Compassion Fatigue Level | At enrollment (single assessment)
  Compassion fatigue will be measured using the Compassion Fatigue Short Scale, which evaluates emotional and physical exhaustion related to caring for individuals experiencing distress. Higher scores indicate greater compassion fatigue.
Work-Related Musculoskeletal Discomfort | Past 7 days
  Work-related musculoskeletal discomfort will be evaluated using the Cornell Musculoskeletal Discomfort Questionnaire, which assesses the frequency, severity, and work interference of musculoskeletal symptoms experienced during the past week.

CONTACTS AND LOCATIONS:
Locations (1):
- Tokat Gaziosmanpaşa University, Faculty of Health Sciences, Tokat Province, Central, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality considerations.

REFERENCES:
- [Background] Devi T., P., Khanwelkar, C., Patil, A., Patil, S. S., Pawar, R., Suruve, D., & Mohana Sundari, S. K. (2019). Compassion Fatigue among Indian Physiotherapists: A descriptive cross sectional comparative study. Global Bioethics Enquiry Journal, 7(1), 17
- [Background] Pena-Curbelo V, Meneses-Monroy A, Mayor-Silva LI, Martin-Casas P, Alvarez-Melcon AC. Work-Related Musculoskeletal Disorders in Physical Therapists: A Cross-Sectional Study. J Clin Med. 2024 Dec 5;13(23):7425. doi: 10.3390/jcm13237425. PMID 39685884
- [Background] Bruschini M, Carli A, Burla F. Burnout and work-related stress in Italian rehabilitation professionals: A comparison of physiotherapists, speech therapists and occupational therapists. Work. 2018;59(1):121-129. doi: 10.3233/WOR-172657. PMID 29439375
- [Background] Tohumcu, K., & Tanrıverdi, D. (2023). The Predictive Effect of Anxiety and Burnout Levels Related to the COVID-19 Pandemic and Organizational Commitment on their Intention to Leave the Organization of the Healthcare Professionals. European Journal of Therapeutics, 29(2), 208-220
- [Background] Yıldız S, Özmenekşe YO. KAÇINILMAZ SON: SESSİZ İSTİFA. Al Farabi Uluslararası Sosyal Bilimler Dergisi. 2024;7(4):14-24.
- [Background] Hedge A, Morimoto S, McCrobie D. Effects of keyboard tray geometry on upper body posture and comfort. Ergonomics. 1999 Oct;42(10):1333-49. doi: 10.1080/001401399184983. PMID 10582503
- [Background] Adams RE, Boscarino JA, Figley CR. Compassion fatigue and psychological distress among social workers: a validation study. Am J Orthopsychiatry. 2006 Jan;76(1):103-8. doi: 10.1037/0002-9432.76.1.103. PMID 16569133